CLINICAL TRIAL: NCT02884960
Title: Safety and Efficacy of Embozene® Microspheres for Uterine Fibroid Embolization Compared to Embosphere® Microspheres for Symptomatic Relief From Uterine Fibroids
Brief Title: Safety and Efficacy of Embozene Microspheres for Uterine Fibroid Embolization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gary Siskin, MD (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Gary Siskin, MD, Professor and Chairman, Department of Radiology, Albany Medical Center, Community Care Physicians, P.C.
Organization: Community Care Physicians, P.C. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1166710
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Uterine Fibroids
Keywords: Uterine Fibroids; Embolization
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Embozene Microspheres (Experimental): Patients will undergo the uterine fibroid embolization procedure with Embozene Microspheres as the embolic agent.
  Interventions: Procedure: Uterine Fibroid Embolization
- Embosphere Microspheres (Active Comparator): Patients will undergo the uterine fibroid embolization procedure with Embosphere Microspheres as the embolic agent.
  Interventions: Procedure: Uterine Fibroid Embolization

INTERVENTIONS:
Procedure: Uterine Fibroid Embolization — This procedure involves the administration of the study device into the uterine arteries to block the flow of blood in these vessels. This deprives fibroid tumors within the uterus of their blood flow, which can cause the tumors to die. This in turn can lead to the relief of symptoms associated with fibroids.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Embozene Microspheres compared with Embosphere Microspheres for the treatment of symptomatic uterine fibroids. A total of 118 patents with symptomatic uterine fibroids will be enrolled at 6 sites. Symptom severity, health-related quality of life, and the appearance of the fibroids will be assessed prior to treatment. Patients will then undergo the uterine fibroid embolization procedure with either Embosphere Microspheres or Embozene Microspheres, which will be randomly assigned. Clinical outcomes will be assessed 1 month, 3 months, 6 months and 12 months after the procedure, and imaging outcomes will be obtained 3 months after the procedure.

DETAILED DESCRIPTION:
The uterine fibroid embolization (UFE) procedure is an accepted, minimally invasive treatment option for patients with symptomatic uterine fibroids. Studies evaluating the outcomes after this procedure have established that the use of polyvinyl alcohol particles and Embosphere Microspheres is associated with best clinical and imaging outcomes. Embozene Microspheres represent a new embolic agent that is being evaluated for use for the treatment of symptomatic fibroids. The purpose of this study is to evaluate the safety and effectiveness of Embozene Microspheres compared with Embosphere Microspheres for the treatment of symptomatic uterine fibroids.

A total of 118 patents with symptomatic uterine fibroids will be enrolled at 6 sites. A questionnaire designed to assess symptom severity and health-related quality of life in patients will be administered to patients at the time of enrollment. In addition, a contrast-enhanced magnetic resonance imaging (MRI) examination will be performed to confirm the diagnosis of fibroids. Patients will then undergo the uterine fibroid embolization procedure. The embolic agent used for the procedure (Embosphere Microspheres or Embozene Microspheres) will be randomly assigned. Patients will be seen 1 month, 3 months, and 6 months and contacted 12 months after the procedure so that the same questionnaire can be used to assess clinical outcomes. In addition, an MRI will be performed 3 months after the procedure to determine the imaging response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. She is able to provide informed consent and sign the Institutional Review Board approved informed consent form.
2. She is pre-menopausal and 30-50 years of age at the time of enrollment.
3. She is not actively attempting to become pregnant for a minimum of 1 year after UFE, or practicing abstinence and willing to continue for a minimum of 1 year after UFE, or is surgically sterile.
4. She is suffering from clinically significant symptoms attributed to the presence of uterine fibroids including abnormal menstrual bleeding and/or bulk-related symptoms including pelvic pain/discomfort, abdominal distension, urinary symptoms (including but not limited to increased urinary frequency or urinary hesitancy), and/or dyspareunia.

Exclusion Criteria:

1. She has a history of pelvic malignancy.
2. She is pregnant or intends to become pregnant within 12 months of the planned UFE procedure.
3. She has had an abnormal PAP smear (anything other than normal or ASCUS - Atypical Squamous Cells of Unknown Significance) within 12 months of the planned UFE procedure.
4. She has a coexisting condition that might explain the presenting symptoms (including but not limited to adenomyosis, endometrial hyperplasia, endometriosis, and complex ovarian cysts).
5. She has evidence of current or recent pelvic inflammatory disease or uterine infection.
6. She has another serious medical condition that might preclude full participation in the study to the desired endpoint (e.g., uncontrolled diabetes, malignancy, chronic obstructive pulmonary disease, myocardial infarction, congestive heart failure, etc.)
7. She has a severe contrast allergy or renal insufficiency that would represent a contraindication to the administration of iodine-based or gadolinium-based contrast agents.
8. She has a contraindication to magnetic resonance imaging (MRI).
9. She has one or more MRI findings including a uterine size >20 cm in greatest length, a dominant fibroid with a greatest diameter >12 cm, an intracavitary submucosal fibroid, or non enhancing dominant fibroids.
10. In the judgment of the investigator, she is unable or unlikely to be able to comply with the study procedures and requirements.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Fibroid Infarction Rate | 3 Months
  The primary effectiveness endpoint for this study is the proportion of patients with a global rate of infarction for all fibroids present within the uterus that is >90% as seen on contrast-enhanced MRI.

SECONDARY OUTCOMES:
Symptom Severity | 12 Months
  The percentage of patients experiencing improvement in symptom severity after the uterine fibroid embolization procedure.
Health-Related Quality of Life | 12 Months
  The percentage of patients experiencing improvement in health-related quality of life after the uterine fibroid embolization procedure.
Uterine Volume | 3 Months
  The change in uterine volume as seen on MRI examinations performed 3 months after the embolization procedure.
Dominant Fibroid Volume | 12 Months
  The change in dominant fibroid volume as seen on MRI examinations performed 3 months after the embolization procedure.
Frequency of Adverse Events After Treatment | 12 Months
  The frequency of adverse events occurring after embolization will be monitored and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Siskin, MD, Principal Investigator — Community Care Physicians

IPD SHARING:
Plan to Share IPD: No